CLINICAL TRIAL: NCT01958021
Title: A Randomized Double-blind, Placebo-controlled Study of LEE011 in Combination With Letrozole for the Treatment of Postmenopausal Women With Hormone Receptor Positive, HER2 Negative, Advanced Breast Cancer Who Received no Prior Therapy for Advanced Disease
Brief Title: Study of Efficacy and Safety of LEE011 in Postmenopausal Women With Advanced Breast Cancer
Acronym: MONALEESA-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEE011A2301; 2013-003084-61 (EudraCT Number)
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Advanced, Metastatic Breast Cancer
Keywords: HR-positive; HER2-negative; Advanced breast cancer; LEE011; Letrozole; CDK; CDK4; CDK6; CDK4/6; Phase III; ER-positive; PR-positive; Postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ribociclib+ letrozole (Experimental): Ribociclib 600 mg daily oral (3 weeks on/ 1 week off) in combination with letrozole 2.5 mg daily oral
  Interventions: Drug: Ribociclib; Drug: Letrozole
- Placebo + letrozole (Placebo Comparator): Placebo daily oral (3 weeks on/ 1 week off) in combination with letrozole 2.5 mg daily oral.
  Participants were unblinded once the final OS analysis was completed and after the implementation of protocol amendment 10 (30-Apr-21) and were given the option to crossover to treatment with ribociclib + letrozole
  Interventions: Drug: Letrozole; Drug: Placebo

INTERVENTIONS:
Drug: Ribociclib — Ribociclib (600 mg, in three 200 mg hard gelatin capsules or tablets) was administered orally once daily on Days 1-21 of each 28-day cycle.
  Other Names: LEE011
  Arms: Ribociclib+ letrozole
Drug: Letrozole — Letrozole (2.5 mg, tablets) was administered orally once daily on a continuous daily schedule (days 1-28 of each 28-day cycle)
Drug: Placebo — Placebo (hard gelatin capsules or tablets) was administered orally once daily on Days 1-21 of each 28-day cycle.
  Arms: Placebo + letrozole

SUMMARY:
The primary purpose of this study was to assess the efficacy of ribociclib, as measured by progression free survival (PFS), in postmenopausal women with hormone receptor positive (HR+), human epidermal growth factor receptor 2 negative (HER2-) advanced breast cancer who received no prior treatment for advanced disease.

DETAILED DESCRIPTION:
This was an international, multi-center, randomized, double-blinded, placebo controlled Phase III trial to determine the efficacy and safety of treatment with ribociclib plus letrozole versus placebo plus letrozole in postmenopausal women with HR+, HER2-negative advanced breast cancer who received no prior therapy for advanced disease.

Eligible patients were randomized in 1:1 ratio to either ribociclib group or placebo group. Study treatment continued until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.

Participants who discontinued treatment due to reasons other than disease progression or withdrawal of consent for efficacy follow-up continued to be monitored until disease progression, death, withdrawal of consent, loss to follow-up, or subject/guardian decision (post-treatment efficacy follow-up).

All participants who discontinued treatment were followed for survival until the predetermined number of overall survival (OS) events was reached.

Following the final OS analysis (performed when approximately 400 deaths were recorded) and with protocol amendment 10 (dated 30-Apr-2021), participants and investigators were unblinded and those participants in the placebo arm had the opportunity to cross-over to the ribociclib arm to receive ribociclib plus letrozole. Cross-over was optional and was conducted at the investigator's discretion and upon participant consent.

ELIGIBILITY:
Key Inclusion Criteria:

1. Women with advanced (locoregionally recurrent or metastatic) breast cancer that was not amenable to curative therapy.
2. The patient was postmenopausal. Postmenopausal status was defined either by:

   * Prior bilateral oophorectomy
   * Age ≥60
   * Age <60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifen, or ovarian suppression) and FSH and estradiol in the postmenopausal range per local normal range.
3. There was no prior systemic anti-cancer therapy for advanced disease.
4. The patient had a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer by the local laboratory.
5. The patient had HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC was 2+, a negative in situ hybridization (FISH, CISH, or SISH) test was required by local laboratory testing.
6. The patient must have had either:

   Measurable disease, i.e., at least one measurable lesion as per RECIST 1.1 criteria (Tumor lesions previously irradiated or subjected to other locoregional therapy were considered measurable if disease progression at the treated site after completion of therapy was clearly documented). OR If no measurable disease was present, then at least one predominantly lytic bone lesion must have been present (Patients with no measurable disease and only one predominantly lytic bone lesion previously irradiated were eligible if there was documented evidence of disease progression of the bone lesion after irradiation).
7. The patient had an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Key Exclusion Criteria:

1. The patient had received any CDK4/6 inhibitor.
2. The patient had received any prior systemic anti-cancer therapy (including hormonal therapy and chemotherapy) for advanced breast cancer.

   Note:
   * Patients who had received (neo) adjuvant therapy for breast cancer were eligible. If the prior neo (adjuvant) therapy included letrozole or anastrozole, the disease-free interval had to be greater than 12 months from the completion of treatment until randomization.
   * Patients who had received ≤ 14 days of letrozole or anastrozole for advanced disease prior to randomization were eligible.
   * Any prior (neo) adjuvant anti-cancer therapy had to be stopped at least 5 half-lives or 7 days, whichever was longer, before randomization.
3. The patient was concurrently using other anti-cancer therapy.
4. The patient had a concurrent malignancy or malignancy within 3 years of randomization, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer, or curatively resected cervical cancer.
5. The patient had active cardiac disease or a history of cardiac dysfunction, including any of the following:

   * History of angina pectoris, symptomatic pericarditis, or myocardial infarction within 12 months prior to study entry.
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV).
   * Documented cardiomyopathy.
   * The patient had a Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO).
   * History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months.
   * On screening, any of the following cardiac parameters: bradycardia (heart rate < 50 at rest), tachycardia (heart rate > 90 at rest), PR interval > 220 msec, QRS interval >109 msec, or QTcF >450 msec.
   * Systolic blood pressure >160 or <90 mmHg.
6. The patient was currently receiving any of the following medications and could not be discontinued 7 days prior to the start of treatment:

   * Medications known to be strong inducers or inhibitors of CYP3A4.
   * Medications known to have a risk of prolonging the QT interval or inducing Torsades de Pointes.
   * Medications with a narrow therapeutic window and predominantly metabolized through CYP3A4.
   * Herbal preparations/medications.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2013-12-17 (Actual); Primary Completion 2016-01-29 (Actual); Study Completion 2023-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (208):
- United States (73):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Arizona Oncology Associates PC HAL, Sedona, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - NEA Baptist Cancer Center, Jonesboro, Arkansas
  - Alta Bates Cancer Center, Berkeley, California
  - City of Hope National Medical Center, Duarte, California
  - Glendale Adventist Medical Center, Glendale, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Cedars Sinai Medical Center SC-5, Los Angeles, California
  - Comprehensive Cancer Center, Sacramento, California
  - Univ of Colorado School of Medicine, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - University Cancer Institute, Boynton Beach, Florida
  - Florida Cancer Research Institute, Davie, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Hospital, Hollywood, Florida
  - University Of Miami, Miami, Florida
  - Florida Retina Institute, Orlando, Florida
  - Sacred Heart Medical Oncology, Pensacola, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Georgia Cancer Specialists, Decatur, Georgia
  - Lewis Hall Singletary Onc Ctr at John D. Archbold Mem Hosp., Thomasville, Georgia
  - Moanalua Medical Center Attn Oncology Dept, Honolulu, Hawaii
  - University of Illinois Cancer Center at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Edward Hospital, Naperville, Illinois
  - IU Simon Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel CCC At JH, Baltimore, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Allina Hlth Cancer Inst Minneapolis, Minneapolis, Minnesota
  - Jackson Oncology Associates, Jackson, Mississippi
  - St Lukes Hos Marion Bloch Neur Inst, Kansas City, Missouri
  - Mercy Medical Research Institute, Manchester, Missouri
  - Foundation Medical Partners, Nashua, New Hampshire
  - Cooper Cancer Center, Camden, New Jersey
  - Hackensack Meridian Health, Edison, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - C R Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Winthrop University Hospital, Mineola, New York
  - NYU Langone Med Center CV Research, New York, New York
  - Mount Sinai School Of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke Univ Medical Center, Durham, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mercy Clinic Oklahoma Communities Mercy Oncology, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Avera Cancer, Sioux Falls, South Dakota
  - Chattanooga Onc And Hem Assoc PC, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Ctr, Nashville, Tennessee
  - Texas Oncology P A, Bedford, Texas
  - Texas Oncology, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Ctr For Cancer And Blood Disorders, Fort Worth, Texas
  - Texas Oncology P A, Fort Worth, Texas
  - Texas Oncology Houston Memorial City, Houston, Texas
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
  - Millennium Research Clin Develop, Houston, Texas
  - Texas Oncology, McAllen, Texas
  - Richardson Hematology Oncology Associates, Richardson, Texas
  - Texas Oncology P A, San Antonio, Texas
  - Texas Oncology Northeast Texas, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia Inc, Salem, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Northwest Medical Specialties, Tacoma, Washington
  - Dean Health System, Madison, Wisconsin
- Argentina (3):
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, La Rioja
- Australia (3):
  - Novartis Investigative Site, Kurralta Park, South Australia
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (5):
  - Novartis Investigative Site, Sint-Niklaas, Oost Vlaanderen
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Wilrijk
- Brazil (2):
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (8):
  - Novartis Investigative Site, Burnaby, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Czechia (4):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Brno-Bohunice
  - Novartis Investigative Site, Liberec
  - Novartis Investigative Site, Olomouc
- Denmark (4):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Odense C
  - Novartis Investigative Site, Vejle
- Finland (2):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Turku
- France (12):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Villejuif
- Germany (19):
  - Novartis Investigative Site, Bielefeld, North Rhine-Westphalia
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Fürth
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Velbert
- Hungary (4):
  - Novartis Investigative Site, Budapest, Pest County
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Gyula
- Ireland (2):
  - Novartis Investigative Site, Cork
  - Novartis Investigative Site, Dublin
- Israel (3):
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (15):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Lecco, LC
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Viterbo, VT
  - Novartis Investigative Site, Napoli
- Lebanon (3):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Netherlands (9):
  - Novartis Investigative Site, Sittard-Geleen, BG
  - Novartis Investigative Site, Leiden, South Holland
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Tilburg
  - Novartis Investigative Site, Zoetermeer
  - Novartis Investigative Site, Zwolle
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
- Russia (3):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Ryazan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Pretoria, Gauteng, South Africa
- South Korea (3):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul
- Spain (8):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Sweden (6):
  - Novartis Investigative Site, Eskilstuna
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Jönköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Uppsala
  - Novartis Investigative Site, Vaxjo
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Diyarbakır
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (2):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Jhaveri K, O'Shaughnessy J, Fasching PA, Tolaney SM, Yardley DA, Sharma VK, Biswas C, Thuerigen A, Pathak P, Rugo HS. Matching-adjusted indirect comparison of PFS and OS comparing ribociclib plus letrozole versus palbociclib plus letrozole as first-line treatment of HR+/HER2- advanced breast cancer. Ther Adv Med Oncol. 2023 Dec 14;15:17588359231216095. doi: 10.1177/17588359231216095. eCollection 2023. PMID 38107828
- [Derived] Andre F, Su F, Solovieff N, Hortobagyi G, Chia S, Neven P, Bardia A, Tripathy D, Lu YS, Lteif A, Taran T, Babbar N, Slamon D, Arteaga CL. Pooled ctDNA analysis of MONALEESA phase III advanced breast cancer trials. Ann Oncol. 2023 Nov;34(11):1003-1014. doi: 10.1016/j.annonc.2023.08.011. Epub 2023 Sep 5. PMID 37673211
- [Derived] Rugo HS, Harmer V, O'Shaughnessy J, Jhaveri K, Tolaney SM, Cardoso F, Bardia A, Maheshwari VK, Tripathi S, Haftchenary S, Pathak P, Fasching PA. Quality of life with ribociclib versus abemaciclib as first-line treatment of HR+/HER2- advanced breast cancer: a matching-adjusted indirect comparison. Ther Adv Med Oncol. 2023 Feb 24;15:17588359231152843. doi: 10.1177/17588359231152843. eCollection 2023. PMID 36861085
- [Derived] Ji Y, Yartsev V, Quinlan M, Serra P, Wang Y, Chakraborty A, Miller M. Justifying Ribociclib Dose in Patients with Advanced Breast Cancer with Renal Impairment Based on PK, Safety, and Efficacy Data: An Innovative Approach Integrating Data from a Dedicated Renal Impairment Study and Oncology Clinical Trials. Clin Pharmacokinet. 2023 Mar;62(3):493-504. doi: 10.1007/s40262-022-01206-2. Epub 2023 Feb 17. PMID 36800111
- [Derived] Hortobagyi GN, Stemmer SM, Burris HA, Yap YS, Sonke GS, Hart L, Campone M, Petrakova K, Winer EP, Janni W, Conte P, Cameron DA, Andre F, Arteaga CL, Zarate JP, Chakravartty A, Taran T, Le Gac F, Serra P, O'Shaughnessy J. Overall Survival with Ribociclib plus Letrozole in Advanced Breast Cancer. N Engl J Med. 2022 Mar 10;386(10):942-950. doi: 10.1056/NEJMoa2114663. PMID 35263519
- [Derived] Burris HA, Chan A, Bardia A, Thaddeus Beck J, Sohn J, Neven P, Tripathy D, Im SA, Chia S, Esteva FJ, Hart L, Zarate JP, Ridolfi A, Lorenc KR, Yardley DA. Safety and impact of dose reductions on efficacy in the randomised MONALEESA-2, -3 and -7 trials in hormone receptor-positive, HER2-negative advanced breast cancer. Br J Cancer. 2021 Aug;125(5):679-686. doi: 10.1038/s41416-021-01415-9. Epub 2021 Jun 22. PMID 34158598
- [Derived] Prat A, Chaudhury A, Solovieff N, Pare L, Martinez D, Chic N, Martinez-Saez O, Braso-Maristany F, Lteif A, Taran T, Babbar N, Su F. Correlative Biomarker Analysis of Intrinsic Subtypes and Efficacy Across the MONALEESA Phase III Studies. J Clin Oncol. 2021 May 1;39(13):1458-1467. doi: 10.1200/JCO.20.02977. Epub 2021 Mar 26. PMID 33769862
- [Derived] Yardley DA. MONALEESA clinical program: a review of ribociclib use in different clinical settings. Future Oncol. 2019 Aug;15(23):2673-2686. doi: 10.2217/fon-2019-0130. Epub 2019 Jul 15. PMID 31305131
- [Derived] Hortobagyi GN. Ribociclib for the first-line treatment of advanced hormone receptor-positive breast cancer: a review of subgroup analyses from the MONALEESA-2 trial. Breast Cancer Res. 2018 Oct 19;20(1):123. doi: 10.1186/s13058-018-1050-7. PMID 30340505
- [Derived] Hortobagyi GN, Stemmer SM, Burris HA, Yap YS, Sonke GS, Paluch-Shimon S, Campone M, Petrakova K, Blackwell KL, Winer EP, Janni W, Verma S, Conte P, Arteaga CL, Cameron DA, Mondal S, Su F, Miller M, Elmeliegy M, Germa C, O'Shaughnessy J. Updated results from MONALEESA-2, a phase III trial of first-line ribociclib plus letrozole versus placebo plus letrozole in hormone receptor-positive, HER2-negative advanced breast cancer. Ann Oncol. 2018 Jul 1;29(7):1541-1547. doi: 10.1093/annonc/mdy155. PMID 29718092
- [Derived] Janni W, Alba E, Bachelot T, Diab S, Gil-Gil M, Beck TJ, Ryvo L, Lopez R, Tsai M, Esteva FJ, Aunon PZ, Kral Z, Ward P, Richards P, Pluard TJ, Sutradhar S, Miller M, Campone M. First-line ribociclib plus letrozole in postmenopausal women with HR+ , HER2- advanced breast cancer: Tumor response and pain reduction in the phase 3 MONALEESA-2 trial. Breast Cancer Res Treat. 2018 Jun;169(3):469-479. doi: 10.1007/s10549-017-4658-x. Epub 2018 Feb 5. PMID 29404806
- [Derived] Hortobagyi GN, Stemmer SM, Burris HA, Yap YS, Sonke GS, Paluch-Shimon S, Campone M, Blackwell KL, Andre F, Winer EP, Janni W, Verma S, Conte P, Arteaga CL, Cameron DA, Petrakova K, Hart LL, Villanueva C, Chan A, Jakobsen E, Nusch A, Burdaeva O, Grischke EM, Alba E, Wist E, Marschner N, Favret AM, Yardley D, Bachelot T, Tseng LM, Blau S, Xuan F, Souami F, Miller M, Germa C, Hirawat S, O'Shaughnessy J. Ribociclib as First-Line Therapy for HR-Positive, Advanced Breast Cancer. N Engl J Med. 2016 Nov 3;375(18):1738-1748. doi: 10.1056/NEJMoa1609709. Epub 2016 Oct 7. PMID 27717303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 223 sites across 29 countries.
Pre-assignment Details: Screening assessments were conducted up to 21 days prior to the randomization
Groups:
- Ribociclib + Letrozole: Ribociclib 600 mg daily oral (3 weeks on/ 1 week off) in combination with letrozole 2.5 mg daily oral
Period: Treatment
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole
Started | 334 | 334
Treated | 334 | 330
Crossover Cohort (Participants in the placebo arm who crossed over to the ribociclib arm and received at least one dose of ribociclib) | 0 | 4
Completed | 0 | 0
Not Completed | 334 | 334
Not completed — Progressive disease | 206 | 265
Not completed — Adverse Event | 38 | 10
Not completed — Subject/guardian decision | 29 | 25
Not completed — Physician Decision | 28 | 21
Not completed — Death | 6 | 1
Not completed — Protocol deviation | 3 | 1
Not completed — Sponsor decision | 24 | 11
Period: Post-treatment Efficacy Follow-up
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole
Started (Patients who discontinue treatment for reasons other than disease progression entered the post-treatment efficacy follow-up. period.) | 26 | 9
Completed | 1 | 0
Not Completed | 25 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Progressive disease | 12 | 3
Not completed — Sponsor decision | 5 | 2
Not completed — Subject/Guardian decision | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole | Total
Number analyzed (Participants) | 334 | 334 | 668
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (10.98) | 61.9 (10.52) | 61.6 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 334 | 334 | 668
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 269 | 280 | 549
  Asian | 28 | 23 | 51
  Black | 10 | 7 | 17
  Native American | 1 | 0 | 1
  Pacific Islander | 1 | 0 | 1
  Other | 12 | 8 | 20
  Unknown | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Investigator Assessment
Description: PFS was defined as the period starting from the date of randomization to the date of the first documented progression or death caused by any reason. In cases where patients did not experience an event, the PFS was censored at the date of the last adequate tumor assessment. Clinical deterioration without objective radiological evidence was not considered as documented disease progression.PFS was assessed by investigator assessment according to RECIST 1.1. The Kaplan-Meier method was used to estimate PFS, and the median PFS, along with 95% confidence intervals, was reported for each treatment group. A stratified Cox regression model was used to estimate the hazard ratio of PFS, along with 95% confidence interval
Time Frame: Up to 23 months
Population: Full Analysis Set (FAS) including all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 334 | 334
months | NA [19.3 to NA] — NA = not estimable due to the insufficient number of participants with events | 14.7 [13.0 to 16.5]
Statistical Analysis 1: Comparison: Ribociclib + Letrozole vs Placebo + Letrozole; Test type: Superiority or Other; p = 0.00000329, Log Rank; Hazard Ratio (HR) = 0.556, 95% CI 2-sided [0.429 to 0.720]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. In cases where the patient's death was not recorded, the OS value was censored at the date of the last known patient's survival status.OS was estimated using the Kaplan-Meier method. As per protocol, the final OS analysis was conducted after approximately 400 deaths were documented.
  The median OS, along with 95% confidence intervals, was reported for each treatment group.The distribution of OS between the two treatment arms was compared using a log-rank test at one-sided cumulative 2.5% level of significance. A stratified Cox regression was used to estimate the OS hazard ratio and the associated 95% CI.
Time Frame: Up to approximately 87 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 334 | 334
Months | 63.9 [52.4 to 71.0] | 51.4 [47.2 to 59.7]
Statistical Analysis 1: Comparison: Ribociclib + Letrozole vs Placebo + Letrozole; Test type: Superiority; p = 0.004, Log Rank; Hazard Ratio (HR) = 0.765, 95% CI 2-sided [0.628 to 0.932]

3. Secondary Outcome: Overall Response Rate (ORR) by Investigator Assessment
Description: ORR is the percentage of participants with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1 as per investigator assessment. . CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 23 months
Population: FAS including all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 334 | 334
Percentage of participants | 40.7 [35.4 to 46.0] | 27.5 [22.8 to 32.3]
Statistical Analysis 1: Comparison: Ribociclib + Letrozole vs Placebo + Letrozole; Test type: Superiority or Other; p = 0.000155, Cochran-Mantel-Haenszel

4. Secondary Outcome: Clinical Benefit Rate (CBR) by Investigator Assessment
Description: Percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD) lasting 24 weeks or longer as defined in RECIST 1.1 as per investigator assessment. CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD = Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease: PD = At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20% the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 23 months
Population: FAS including all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 334 | 334
Percentage of participants | 79.6 [75.3 to 84.0] | 72.8 [68.0 to 77.5]
Statistical Analysis 1: Comparison: Ribociclib + Letrozole vs Placebo + Letrozole; Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel

5. Secondary Outcome: Time to Definitive Deterioration of Eastern Cooperative Oncology Group Performance Status (ECOG PS) by at Least One Category of the Score
Description: ECOG PS categorized patients based on their ability to perform daily activities and self-care, with scores ranging from 0 to 5. A score of 0 indicated no restrictions in activity, while higher scores indicated increasing limitations. Time to definitive deterioration was defined as the time from the date of randomization to the date of the event, defined as experiencing an increase in ECOG PS by at least one category from the baseline or death. A deterioration was considered definitive if no improvements in the ECOG PS were observed at a subsequent time. The Kaplan-Meier method was used to estimate the distribution, and the median time to definitive deterioration, along with 95% confidence intervals, was reported for each treatment group. Patients receiving any further therapy prior to definitive worsening were censored at their date of last assessment prior to start of therapy. Patients that had not worsened at the data cutoff point were censored at the date of last assessment.
Time Frame: From baseline up to 23 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 334 | 334
Months | 22.6 [22.6 to NA] — NA= Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA= Not estimable due to the insufficient number of participants with events

6. Secondary Outcome: Time to Definitive 10% Deterioration in the Global Health Status/Quality of Life (GHS/QoL) Scale Score of the European Organization for Research and Treatment of Cancer's Core Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 is a questionnaire that includes 5 functional scales, 3 symptom scales, 1 GHS/QoL scale, and 6 single items. GHS/QoL scale score ranges between 0 and 100. A high score for GHS/QoL represents better functioning or QoL.The time to definitive 10% deterioration is defined as the time from the date of randomization to the date of event, which is defined as at least 10% relative to baseline worsening of the QoL score (without further improvement above the threshold) or death due to any cause. The Kaplan-Meier method was used to estimate the distribution, and the median time to definitive 10% deterioration, along with 95% confidence intervals, was reported for each treatment group. If a patient had not had an event, time to deterioration was censored at the date of the last adequate QoL evaluation.
Time Frame: From baseline up to 23 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 334 | 334
Months | 19.3 [16.6 to 22.1] | NA [14.8 to NA] — NA= Not estimable due to the insufficient number of participants with events

7. Secondary Outcome: Change From Baseline in the GHS/QoL Scale Score of the EORTC QLQ-C30
Description: The EORTC QLQ-C30 is a questionnaire that includes 5 functional scales, 3 symptom scales, 1 GHS/QoL scale, and 6 single items. GHS/QoL scale score ranges between 0 and 100. A high score for GHS/QoL represents better functioning or QoL.The change from baseline in the GHS/QoL score was assesed. A positive change from baseline indicated improvement.
  For subjects who discontinued treatment earlier and without disease progression, post-treatment efficacy follow-up visits occurred every 8 weeks after End of treatment (EOT) during the initial 18 months since start of treatment, followed by visits every 12 weeks until disease progression or end of study.
Time Frame: Baseline, every 2 cycles for 18 months, then every 3 cycles until last dose; at EOT (within 15 days from last dose);every 8 or 12 weeks post-treatment until progression (post-treatment efficacy visits), assessed up to 23 months. Cycle=28 days
Population: Randomized participants with data available at the specified time points. Number analyzed refers to the number of participants with an evaluable value at the specified time point.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 285 | 285
Score on a Scale
  Cycle 3 Day 1 | 2.9 (18.68) | 4.9 (19.14)
  Cycle 5 Day 1: number analyzed (Participants) | 262 | 254
  Cycle 5 Day 1 | 4.6 (19.86) | 6.8 (19.64)
  Cycle 7 Day 1: number analyzed (Participants) | 249 | 248
  Cycle 7 Day 1 | 4.6 (20.96) | 6.0 (20.19)
  Cycle 9 Day 1: number analyzed (Participants) | 232 | 219
  Cycle 9 Day 1 | 5.1 (21.95) | 8.0 (20.49)
  Cycle 11 Day 1: number analyzed (Participants) | 223 | 193
  Cycle 11 Day 1 | 4.9 (21.11) | 7.0 (20.45)
  Cycle 13 Day 1: number analyzed (Participants) | 203 | 177
  Cycle 13 Day 1 | 5.3 (22.37) | 6.5 (20.40)
  Cycle 15 Day 1: number analyzed (Participants) | 152 | 129
  Cycle 15 Day 1 | 5.5 (21.43) | 8.7 (21.23)
  Cycle 17 Day 1: number analyzed (Participants) | 108 | 80
  Cycle 17 Day 1 | 4.6 (22.85) | 7.4 (21.75)
  Cycle 19 Day 1: number analyzed (Participants) | 60 | 40
  Cycle 19 Day 1 | 5.0 (23.08) | 7.7 (18.81)
  Cycle 22 Day 1: number analyzed (Participants) | 19 | 14
  Cycle 22 Day 1 | 4.8 (20.09) | 12.5 (14.15)
  Cycle 25 Day 1: number analyzed (Participants) | 3 | 0
  Cycle 25 Day 1 | -8.3 (8.33) |
  EOT: number analyzed (Participants) | 97 | 142
  EOT | -1.2 (20.97) | -1.2 (15.30)
  Post -treatment efficacy visit 1: number analyzed (Participants) | 4 | 3
  Post -treatment efficacy visit 1 | 8.3 (28.87) | -16.7 (16.67)
  Post -treatment efficacy visit 2: number analyzed (Participants) | 7 | 2
  Post -treatment efficacy visit 2 | 3.6 (17.25) | -20.8 (17.68)
  Post -treatment efficacy visit 3: number analyzed (Participants) | 5 | 2
  Post -treatment efficacy visit 3 | 5.0 (21.73) | -12.5 (5.89)
  Post -treatment efficacy visit 4: number analyzed (Participants) | 4 | 2
  Post -treatment efficacy visit 4 | 6.3 (28.36) | 8.3 (0.00)
  Post -treatment efficacy visit 5: number analyzed (Participants) | 3 | 2
  Post -treatment efficacy visit 5 | 0.0 (28.87) | -4.2 (5.89)
  Post -treatment efficacy visit 6: number analyzed (Participants) | 2 | 0
  Post -treatment efficacy visit 6 | 20.8 (41.25) |
  Post -treatment efficacy visit 7: number analyzed (Participants) | 1 | 0
  Post -treatment efficacy visit 7 | 50.0 |

8. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from randomization to the day before first dose of study medication.
  On-treatment deaths were collected from start of treatment to 30 days after last dose of treatment or one day before first administration of crossover treatment (for crossover participants), whichever came first Crossover on-treatment deaths were collected from start of crossover treatment up to 30 days after last dose of crossover treatment.
  Post-treatment survival follow-up (FU) deaths were collected from day 31 after last dose of study treatment to end of study.
  Crossover post-treatment survival FU deaths were collected from day 31 after last dose of crossover treatment to end of study
Time Frame: Pre-treatment: Up to 21 days. On-treatment: Up to 99 months. Crossover on-treatment: Up to 12 months after crossing-over.Post-treatment survival FU: Up to 99 months.Crossover post-treatment survival FU: Up to 12 months after crossing-over
Population: FAS including all randomized participants
Measure: Number; unit: Participants
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 334 | 334
Participants
  Pre-treatment | 0 | 0
  On-treatment: number analyzed (Participants) | 334 | 330
  On-treatment | 8 | 3
  Crossover On-treatment: number analyzed (Participants) | 0 | 4
  Crossover On-treatment |  | 0
  Post-treatment survival follow-up: number analyzed (Participants) | 278 | 298
  Post-treatment survival follow-up | 178 | 218
  Crossover post-treatment survival follow-up: number analyzed (Participants) | 0 | 4
  Crossover post-treatment survival follow-up |  | 0
  All deaths | 186 | 221

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM): from randomization up to 99 months, including post-treatment survival follow-up (FU). If crossover, ACM also collected from start of crossover treatment to 12 months, including post-treatment survival FU. Serious and Other Adverse Events (AEs): from 1st dose of treatment to 30 days after last dose (or start of crossover treatment), up to 99 months. If crossover, AEs also collected from start of crossover treatment to 30 days post-crossover treatment, up to 12 months
Description: All-cause mortality: reported for all randomized participants regardless of whether the assigned study treatment was received. Deaths in post-treatment survival follow-up period (more than 30 days after last dose) are reported separately and are not considered AEs.
  Serious and Other AEs: reported for all randomized participants who received at least one dose of study treatment
Groups:
- Ribociclib + Letrozole: All-cause mortality from randomization until 30 days after last dose. Adverse Events from first dose until 30 days after last dose.
- Placebo + Letrozole: All-cause mortality from randomization until 30 days after last dose or start of crossover treatment. Adverse Events from first dose until 30 days after last dose or start of crossover treatment.
- Crossover to Ribociclib + Letrozole: All-cause mortality and Adverse Events from start of crossover treatment to 30 days post-crossover treatment
- Ribociclib + Letrozole (Post-treatment Survival Follow-up); Placebo + Letrozole (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 after last dose). No AEs were collected during this period
- Crossover to Ribociclib + Fulvestrant (Crossover Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 after last dose of crossover treatment). No AEs were collected during this period
Arm/Group | Ribociclib + Letrozole | Placebo + Letrozole | Crossover to Ribociclib + Letrozole | Ribociclib + Letrozole (Post-treatment Survival Follow-up) | Placebo + Letrozole (Post-treatment Survival Follow-up) | Crossover to Ribociclib + Fulvestrant (Crossover Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 8/334 | 3/334 | 0/4 | 178/278 | 218/298 | 0/4
Serious Adverse Events (participants affected / at risk) | 108/334 | 62/330 | 1/4 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 331/334 | 317/330 | 4/4 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib + Letrozole (N=334) | Placebo + Letrozole (N=330) | Crossover to Ribociclib + Letrozole (N=4) | Ribociclib + Letrozole (Post-treatment Survival Follow-up) (N=0) | Placebo + Letrozole (Post-treatment Survival Follow-up) (N=0) | Crossover to Ribociclib + Fulvestrant (Crossover Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 0 | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | NA | NA | NA
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | NA | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | NA | NA | NA
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | NA | NA | NA
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Cor pulmonale (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Coronary artery disease (Cardiac disorders) | 0 | 2 | 0 | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | NA | NA | NA
Cataract (Eye disorders) | 1 | 2 | 0 | NA | NA | NA
Glaucoma (Eye disorders) | 0 | 1 | 0 | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 6 | 0 | 0 | NA | NA | NA
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | NA | NA | NA
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 4 | 0 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | NA | NA | NA
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | NA | NA | NA
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 5 | 2 | 0 | NA | NA | NA
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0 | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 5 | 3 | 0 | NA | NA | NA
Asthenia (General disorders) | 1 | 0 | 0 | NA | NA | NA
Chest discomfort (General disorders) | 0 | 1 | 0 | NA | NA | NA
General physical health deterioration (General disorders) | 5 | 2 | 0 | NA | NA | NA
Malaise (General disorders) | 1 | 0 | 0 | NA | NA | NA
Non-cardiac chest pain (General disorders) | 3 | 1 | 0 | NA | NA | NA
Oedema peripheral (General disorders) | 2 | 0 | 0 | NA | NA | NA
Pyrexia (General disorders) | 2 | 1 | 0 | NA | NA | NA
Sudden death (General disorders) | 1 | 0 | 0 | NA | NA | NA
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0 | NA | NA | NA
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 2 | 1 | 0 | NA | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 3 | 0 | 0 | NA | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | NA | NA | NA
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Abscess jaw (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Bronchitis (Infections and infestations) | 1 | 1 | 0 | NA | NA | NA
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Cellulitis (Infections and infestations) | 2 | 1 | 0 | NA | NA | NA
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Diverticulitis (Infections and infestations) | 1 | 1 | 0 | NA | NA | NA
Encephalitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Erysipelas (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Pneumonia (Infections and infestations) | 8 | 3 | 0 | NA | NA | NA
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Retroperitoneal abscess (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Sepsis (Infections and infestations) | 3 | 1 | 0 | NA | NA | NA
Skin infection (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | NA | NA | NA
Urosepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Wound infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | NA | NA | NA
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | NA | NA | NA
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | NA | NA | NA
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | NA | NA | NA
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 4 | 0 | 0 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0 | NA | NA | NA
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Blood creatinine increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1 | 0 | NA | NA | NA
C-reactive protein increased (Investigations) | 0 | 1 | 0 | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | NA | NA | NA
International normalised ratio increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Waist circumference increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Weight decreased (Investigations) | 1 | 0 | 0 | NA | NA | NA
White blood cell count decreased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 4 | 2 | 0 | NA | NA | NA
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | NA | NA | NA
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA | NA | NA
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | NA | NA | NA
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA | NA | NA
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | 5 | 2 | 0 | NA | NA | NA
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 0 | 3 | 0 | NA | NA | NA
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Migraine (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Presyncope (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Spinal cord compression (Nervous system disorders) | 2 | 1 | 0 | NA | NA | NA
Syncope (Nervous system disorders) | 4 | 2 | 0 | NA | NA | NA
Toxic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | NA | NA | NA
Major depression (Psychiatric disorders) | 1 | 0 | 0 | NA | NA | NA
Mental status changes (Psychiatric disorders) | 2 | 1 | 0 | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 0 | NA | NA | NA
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Renal failure (Renal and urinary disorders) | 2 | 2 | 0 | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | NA | NA | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 0 | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | NA | NA | NA
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | NA | NA | NA
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Embolism (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Hypertension (Vascular disorders) | 1 | 1 | 0 | NA | NA | NA
Hypotension (Vascular disorders) | 2 | 0 | 0 | NA | NA | NA
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0 | NA | NA | NA
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib + Letrozole (N=334) | Placebo + Letrozole (N=330) | Crossover to Ribociclib + Letrozole (N=4) | Ribociclib + Letrozole (Post-treatment Survival Follow-up) (N=0) | Placebo + Letrozole (Post-treatment Survival Follow-up) (N=0) | Crossover to Ribociclib + Fulvestrant (Crossover Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 77 | 24 | 2 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 56 | 10 | 2 | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 19 | 7 | 1 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 218 | 18 | 2 | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 24 | 3 | 0 | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 27 | 7 | 0 | NA | NA | NA
Dry eye (Eye disorders) | 27 | 13 | 0 | NA | NA | NA
Lacrimation increased (Eye disorders) | 39 | 7 | 0 | NA | NA | NA
Vision blurred (Eye disorders) | 17 | 9 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 41 | 33 | 0 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 31 | 21 | 0 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 99 | 75 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 137 | 88 | 2 | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 48 | 37 | 0 | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 37 | 25 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 183 | 106 | 3 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 53 | 24 | 1 | NA | NA | NA
Toothache (Gastrointestinal disorders) | 18 | 14 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 115 | 62 | 0 | NA | NA | NA
Asthenia (General disorders) | 49 | 49 | 1 | NA | NA | NA
Chest discomfort (General disorders) | 1 | 4 | 1 | NA | NA | NA
Chills (General disorders) | 17 | 11 | 0 | NA | NA | NA
Fatigue (General disorders) | 145 | 119 | 1 | NA | NA | NA
Influenza like illness (General disorders) | 23 | 23 | 1 | NA | NA | NA
Non-cardiac chest pain (General disorders) | 18 | 29 | 0 | NA | NA | NA
Oedema peripheral (General disorders) | 49 | 41 | 0 | NA | NA | NA
Pyrexia (General disorders) | 49 | 24 | 0 | NA | NA | NA
Acarodermatitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Bronchitis (Infections and infestations) | 25 | 18 | 0 | NA | NA | NA
Conjunctivitis (Infections and infestations) | 18 | 5 | 0 | NA | NA | NA
Influenza (Infections and infestations) | 26 | 18 | 0 | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 37 | 29 | 0 | NA | NA | NA
Sinusitis (Infections and infestations) | 22 | 16 | 0 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 51 | 43 | 0 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 53 | 37 | 0 | NA | NA | NA
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 66 | 21 | 1 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 66 | 23 | 1 | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 22 | 21 | 0 | NA | NA | NA
Blood creatinine increased (Investigations) | 37 | 9 | 1 | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 17 | 5 | 0 | NA | NA | NA
Lymphocyte count decreased (Investigations) | 26 | 3 | 1 | NA | NA | NA
Neutrophil count decreased (Investigations) | 78 | 5 | 2 | NA | NA | NA
Platelet count decreased (Investigations) | 11 | 0 | 1 | NA | NA | NA
Weight decreased (Investigations) | 29 | 16 | 1 | NA | NA | NA
White blood cell count decreased (Investigations) | 70 | 8 | 1 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 74 | 61 | 1 | NA | NA | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12 | 10 | 1 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 29 | 25 | 0 | NA | NA | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 17 | 17 | 0 | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 21 | 6 | 0 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 11 | 0 | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 7 | 1 | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 3 | 1 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 135 | 136 | 0 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 91 | 76 | 0 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 44 | 47 | 0 | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26 | 28 | 0 | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 21 | 27 | 0 | NA | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 17 | 0 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 35 | 30 | 0 | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 20 | 21 | 0 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 62 | 63 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | 54 | 53 | 1 | NA | NA | NA
Dysgeusia (Nervous system disorders) | 20 | 14 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 98 | 76 | 1 | NA | NA | NA
Paraesthesia (Nervous system disorders) | 17 | 13 | 0 | NA | NA | NA
Taste disorder (Nervous system disorders) | 17 | 8 | 0 | NA | NA | NA
Anxiety (Psychiatric disorders) | 41 | 29 | 0 | NA | NA | NA
Depression (Psychiatric disorders) | 33 | 29 | 0 | NA | NA | NA
Insomnia (Psychiatric disorders) | 55 | 49 | 0 | NA | NA | NA
Breast pain (Reproductive system and breast disorders) | 21 | 23 | 0 | NA | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 8 | 16 | 1 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 89 | 83 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 | 44 | 0 | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 10 | 0 | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 | 21 | 0 | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 119 | 55 | 0 | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 34 | 12 | 0 | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 23 | 6 | 0 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 61 | 27 | 0 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 68 | 33 | 0 | NA | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | NA | NA | NA
Vitiligo (Skin and subcutaneous tissue disorders) | 6 | 0 | 1 | NA | NA | NA
Hot flush (Vascular disorders) | 84 | 88 | 0 | NA | NA | NA
Hypertension (Vascular disorders) | 71 | 69 | 0 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.